CLINICAL TRIAL: NCT05421624
Title: Amped-PD: Amplifying Physical Activity Through a Novel Digital Music Therapeutic in Parkinson Disease
Brief Title: Amped-PD: Amplifying Physical Activity Through Music in Parkinson Disease
Acronym: Amped-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: University of New England (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6518; P30AG048785 (NIH)
Record Dates: First submitted 2022-06-09; First posted 2022-06-16 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; rhythmic auditory stimulation; digital therapeutics; behavior change; habits; physical activity
MeSH Terms: conditions — Parkinson Disease; Habits; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either intervention of (1) Amped-PD, or (2) Active-Control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Amped-PD (Experimental): 6-week community-based, self-directed walking program that uses a novel digital therapeutic that delivers music-adaptive rhythmic auditory stimulation.
  Interventions: Device: Digital music therapeutic
- Active-Control (Active Comparator): 6-week community-based, self-directed walking program without using a novel digital therapeutic or any form of rhythmic auditory stimulation.
  Interventions: Behavioral: Active-Control

INTERVENTIONS:
Device: Digital music therapeutic — The digital music therapeutic is comprised of foot sensors, a smart phone with pre-installed proprietary software application, and headphones. The device obtains real-time walking data through movement sensors that communicate wirelessly with the smartphone application software. Music cues are tailored to the person's walking pattern, and are transmitted wirelessly to the headphones. Music cues are time-shifted to the user's baseline cadence and adjusted in real-time based on the user's walking performance metrics.
  Other Names: MedRhythms device
  Arms: Amped-PD
Behavioral: Active-Control — The Active-Control intervention will implement a similarly structured community-based walking program as Amped-PD, with the only exception the digital music therapeutic.
  Arms: Active-Control

SUMMARY:
Regular, habitual exercise is a critical component of the long-term management of Parkinson disease (PD). However, PD-specific motor (e.g. slow and diminished movements, variable step timing) and non-motor (e.g. depression, apathy) problems collectively hinder physical activity. Rhythmic auditory stimulation (RAS) is a rehabilitation technique that employs coupling of auditory cues with movement. Walking with RAS has been shown to benefit walking rhythmicity, quality, and speed. These walking benefits make RAS advantageous in promoting moderate intensity walking activity -- an important health-objective in the management of PD. However, the therapeutic potential of RAS in self-directed walking programs has not been examined. In this pilot, we will utilize a breakthrough digital therapeutic that delivers music-adaptive RAS to alleviate PD-specific problems by regulating stepping patterns. Using music as a substrate for cue delivery, this digital therapeutic leverages gait benefits from RAS along with enjoyment of music listening, thus making it a viable and engaging modality that will yield habits of regular walking. Habits are automatically recurring psychological dispositions that emerge from repeated behaviors. The investigators posit that music cues provide recurring contextual cues that automatically evoke habitual response of exercise, thus has the potential to prompt regular physical activity. This study will enroll 61individuals with mild-to-moderate PD (Run-in: 17; Main Trial: 44). The experimental intervention, "Amped-PD", is a 6-week, user-managed community-based walking program that utilizes music-adaptive RAS that progressively increases walking intensities. This study will examine if Amped-PD (Experimental Intervention) is more effective than a standard-of-care walking program (Active-Control Intervention) in improving physical activity based on moderate intensity walking, and in improving motor deficits related to quality of walking in individuals with mild-to-moderate PD. This study will also examine whether the resultant habits formed from each intervention matter in relation to training-related changes in physical activity.

DETAILED DESCRIPTION:
Parkinson disease (PD) is the fastest growing source of disability among neurological disorders. Diminished physical activity is highly prevalent in PD and often lead to the onset of disability. Regular, habitual exercise is a critical component of the long-term PD management. However, PD-specific motor (e.g. slow and diminished movements, variable step timing) and non-motor (e.g. depression, apathy) problems collectively hinder physical activity. Rhythmic auditory stimulation (RAS) is a rehabilitation technique that employs the coupling of auditory cues with movement. When used during walking, RAS has been shown to benefit walking rhythmicity, quality, and speed. Therefore this rehabilitation technique can be advantageous in promoting moderate intensity walking activity. While clinical studies support RAS-based intervention, its translation to real-world, community-based environments and for long-term exercise for the promotion of physical activity is limited. The difference that determines viability of RAS for out-of-lab applications lie in the distinction between external entrainment (open-loop) versus autonomous entrainment (closed-loop). Open-loop RAS requires high levels of vigilance and is prone to error accumulation, which is problematic with gait dysfunction in PD. On the other hand, closed-loop RAS allows for natural and stable entrainment. A closed-loop approach in this case is a necessity of the task and a technological challenge to translate RAS to community-based settings. In this pilot, the investigators will utilize a breakthrough digital therapeutic that employs closed-loop RAS to alleviate PD-specific problems by regulating stepping patterns. Using music as a substrate for cue delivery, this digital therapeutic leverages gait benefits from RAS along with enjoyment of music listening, thus making it a viable and engaging modality that will yield habits of regular walking. The investigators posit that music that is linked to enjoyment serves as context cues that define the pre-condition to engaging in habitual walking exercise and increased physical activity. With repetition, these recurring contextual triggers (i.e. music) automatically evoke a habitual response of exercise, and thus has the potential to amplify physical activity.

The main aims of the study seek to examine if Amped-PD (Experimental Intervention) is more effective than a standard-of-care walking program (Active-Control Intervention) in improving physical activity based on moderate intensity walking (Aim 1), and in improving motor deficits related to quality of walking (Aim 2) in individuals with mild-to-moderate PD. Additionally, this study will examine whether habit formation mediates the relationship between the intervention (Amped-PD or Active-Control) and physical activity (Aim 3). The investigators hypothesize that Amped-PD will have greater improvements in amounts of moderate intensity walking and stride-to-stride variability based on stride length and swing time. Further, habit formation will be one mechanism that will explain the link between the intervention and physical activity. Secondary research aims will examine whether Amped-PD is more effective than Active-Control in improving motor and non-motor features based on short- and long-distance walking function, spatiotemporal measures of walking, step activity based on daily step counts, disease severity scores, quality of life, self-efficacy on walking, and depression.

This study will utilize the breakthrough digital music therapeutic developed and manufactured by MedRhythms (Portland, ME). To examine the effects of the intervention, the investigators will use clinical measures of motor and gait function, participant self-reports on habit formation, and quantified movement data on walking and physical activity using wearable sensors. This study will be implemented by carrying out the following study visits: (1) Primary screen over the phone, (2) Clinical Screening and Baseline Assessment, (3) Community-based, self-directed walking program (6 weeks), (3) Post-training Assessment; (4) Follow-up training (2 weeks), and (5) Final Follow-Up Assessment. Altogether, these procedures may take up to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic, typical Parkinson disease (based on the UK PD Society Brain Bank Criteria7) by a physician
* Modified Hoehn and Yahr stages 1-3 per physical exam by a licensed physical therapist
* 40 - 85 years of age
* Community-dwelling
* Able to walk independently without physical assistance or an assistive device for at least 10 minutes.
* Have stable PD medications for at least two weeks prior to enrollment.
* Willing and able to provide informed consent.
* Provide HIPAA Authorization to allow communication with the primary healthcare provider for communication (as needed) during the study period.

Exclusion Criteria:

* < 40 years of age
* Diagnosis of atypical Parkinsonism
* Modified Hoehn and Yahr stages 4-5
* Moderately or significantly disturbing freezing episodes during daily walking based on the New Freezing of Gait Questionnaire
* History of >1 fall over the past 3 months
* Cognitive impairment (i.e., Mini-Mental State Exam Score (MMSE) < 24)
* Unable to walk independently (i.e. without physical assistance or assistive device) at a comfortable speed of 0.4m/s or greater (i.e., 10-meter Walk Test (10mWT))
* Unable to independently use the music-based digital therapeutic during training
* Significant hearing impairment
* Currently participating in physical therapy
* Currently performing regular walking exercise > 3x/week for 30 minutes per session.
* Cardiac conditions that may limit safe participation in exercise
* Orthopedic conditions that may limit safe participation in exercise
* Any other medical conditions that would preclude successful participation as determined by a physical therapist

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franchino Porciuncula, PT, EdD, Principal Investigator — Boston University; Terry D. Ellis, PT, PhD, Principal Investigator — Boston University
Locations (1):
- Center for Neurorehabilitation at Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavanaugh JT, Ellis TD, Earhart GM, Ford MP, Foreman KB, Dibble LE. Toward Understanding Ambulatory Activity Decline in Parkinson Disease. Phys Ther. 2015 Aug;95(8):1142-50. doi: 10.2522/ptj.20140498. Epub 2015 Apr 9. PMID 25858971
- [Background] Ellis TD, Cavanaugh JT, Earhart GM, Ford MP, Foreman KB, Thackeray A, Thiese MS, Dibble LE. Identifying clinical measures that most accurately reflect the progression of disability in Parkinson disease. Parkinsonism Relat Disord. 2016 Apr;25:65-71. doi: 10.1016/j.parkreldis.2016.02.006. Epub 2016 Feb 2. PMID 26876037
- [Background] Nombela C, Hughes LE, Owen AM, Grahn JA. Into the groove: can rhythm influence Parkinson's disease? Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2564-70. doi: 10.1016/j.neubiorev.2013.08.003. Epub 2013 Sep 3. PMID 24012774
- [Background] Thaut MH, McIntosh GC, Rice RR, Miller RA, Rathbun J, Brault JM. Rhythmic auditory stimulation in gait training for Parkinson's disease patients. Mov Disord. 1996 Mar;11(2):193-200. doi: 10.1002/mds.870110213. PMID 8684391
- [Background] Hutchinson K, Sloutsky R, Collimore A, Adams B, Harris B, Ellis TD, Awad LN. A Music-Based Digital Therapeutic: Proof-of-Concept Automation of a Progressive and Individualized Rhythm-Based Walking Training Program After Stroke. Neurorehabil Neural Repair. 2020 Nov;34(11):986-996. doi: 10.1177/1545968320961114. Epub 2020 Oct 10. PMID 33040685
- [Background] Gardner B. A review and analysis of the use of 'habit' in understanding, predicting and influencing health-related behaviour. Health Psychol Rev. 2015;9(3):277-95. doi: 10.1080/17437199.2013.876238. Epub 2014 Jan 21. PMID 25207647
- [Background] Galla BM, Duckworth AL. More than resisting temptation: Beneficial habits mediate the relationship between self-control and positive life outcomes. J Pers Soc Psychol. 2015 Sep;109(3):508-25. doi: 10.1037/pspp0000026. Epub 2015 Feb 2. PMID 25643222
- [Background] Wittwer JE, Winbolt M, Morris ME. Home-Based Gait Training Using Rhythmic Auditory Cues in Alzheimer's Disease: Feasibility and Outcomes. Front Med (Lausanne). 2020 Jan 31;6:335. doi: 10.3389/fmed.2019.00335. eCollection 2019. PMID 32083083
- [Background] Jeng B, Cederberg KL, Lai B, Sasaki JE, Bamman MM, Motl RW. Step-rate threshold for physical activity intensity in Parkinson's disease. Acta Neurol Scand. 2020 Aug;142(2):145-150. doi: 10.1111/ane.13250. Epub 2020 Apr 22. PMID 32255504
- [Background] Tudor-Locke C, Craig CL, Aoyagi Y, Bell RC, Croteau KA, De Bourdeaudhuij I, Ewald B, Gardner AW, Hatano Y, Lutes LD, Matsudo SM, Ramirez-Marrero FA, Rogers LQ, Rowe DA, Schmidt MD, Tully MA, Blair SN. How many steps/day are enough? For older adults and special populations. Int J Behav Nutr Phys Act. 2011 Jul 28;8:80. doi: 10.1186/1479-5868-8-80. PMID 21798044
- [Derived] Cavanaugh JT, Porciuncula F, Zajac JA, Baker T, Wendel N, Awad LN, Ellis TD. Gait Responses in People with Parkinson Disease During Autonomous Closed-loop Rhythmic Auditory Stimulation: An Exploratory Analysis. Neurorehabil Neural Repair. 2025 Aug;39(8):666-676. doi: 10.1177/15459683251340910. Epub 2025 May 29. PMID 40438970
- [Derived] Porciuncula F, Cavanaugh JT, Zajac J, Wendel N, Baker T, Arumukhom Revi D, Eklund N, Holmes MB, Awad LN, Ellis TD. Amplifying walking activity in Parkinson's disease through autonomous music-based rhythmic auditory stimulation: randomized controlled trial. NPJ Parkinsons Dis. 2025 Apr 29;11(1):100. doi: 10.1038/s41531-025-00952-x. PMID 40301366

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amped-PD | Active-Control
Started | 22 | 22
Completed | 21 | 20
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Participant baseline was based on completer analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amped-PD | Active-Control | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.95 (8.84) | 60.065 (9.13) | 63.87 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 19 | 40
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41
Unified Parkinson's Disease Rating Scale Part III Score [Mean (Standard Deviation); unit: Points] — The MDS UPDRS is the most widely used clinical rating scale for Parkinson disease. Part III is a motor examination (33 scores summed from 18 questions) conducted by the rater. The total score is reported, which can range from 0 (no impairment) to 141 (maximum impairment).
  Points | 20.71 (7.68) | 22.75 (10.60) | 20.73 (8.57)

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Based on the Amount of Moderate Intensity Walking
Description: The amount of moderate intensity walking, defined as mean number of minutes per day with >100 steps/min. This will be measured using research-grade activity monitors (StepWatch Activity Monitor, Modus Health, Edmonds, WA) validated for use in PD.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes of moderate intensity walking
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 16
minutes of moderate intensity walking | 9.45 (9.39) | 16.17 (18.08)

2. Primary Outcome: Physical Activity Based on the Amount of Moderate Intensity Walking
Description: as for outcome 1
Time Frame: During training up to 4 days from start of training
Measure: Mean (Standard Deviation); unit: minutes of moderate intensity walking
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 16
minutes of moderate intensity walking | 32.83 (10.14) | 23.08 (12.09)

3. Primary Outcome: Physical Activity Based on the Amount of Moderate Intensity Walking
Description: as for outcome 1
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: minutes of moderate intensity walking
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 16
minutes of moderate intensity walking | 30.30 (11.45) | 24.15 (15.23)

4. Primary Outcome: Physical Activity Based on the Amount of Moderate Intensity Walking
Description: as for outcome 1
Time Frame: Follow-up (up to 2 weeks post-intervention)
Measure: Mean (Standard Deviation); unit: minutes of moderate intensity walking
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 16
minutes of moderate intensity walking | 6.85 (6.48) | 13.22 (9.62)

5. Primary Outcome: Step Activity Based on Daily Step Counts
Description: Daily step counts refer to the total number of steps taken on the leg with the monitor. This will be measured using research-grade activity monitors (StepWatch Activity Monitor, Modus Health, Edmonds, WA) validated for use in PD.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 16
steps | 8812 (3453) | 10311 (3497)

6. Primary Outcome: Step Activity Based on Daily Step Counts
Description: as for outcome 5
Time Frame: During training up to 4 days from start of training
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 16
steps | 12155 (3127) | 10483 (3751)

7. Primary Outcome: Step Activity Based on Daily Step Counts
Description: as for outcome 5
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 16
steps | 11346 (2665) | 10926 (2756)

8. Primary Outcome: Step Activity Based on Daily Step Counts
Description: as for outcome 5
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 16
steps | 8407 (2967) | 8284 (3933)

9. Primary Outcome: Gait Quality Based on Variability of Stride Time
Description: Stride-to-stride variability of stride time of the gait cycle will be measured using wearable sensors. Stride time variability is calculated by dividing the standard deviation of stride time by the mean of stride time, multiplied by 100 to express as percentage. Worse gait quality is indicated by higher stride time variability, while improved gait quality is indicated by lower stride time variability.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: %coefficient of variation
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 19 | 15
%coefficient of variation | 4.19 (2.38) | 2.88 (0.81)

10. Primary Outcome: Gait Quality Based on Variability of Stride Time
Description: as for outcome 9
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: %coefficient of variation
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 19 | 15
%coefficient of variation | 3.46 (1.64) | 3.18 (1.07)

11. Primary Outcome: Gait Quality Based on Variability of Stride Time
Description: as for outcome 9
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: %coefficient of variation
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 19 | 15
%coefficient of variation | 3.70 (2.01) | 3.05 (1.70)

12. Primary Outcome: Self-Report Habit Index (SRHI)
Description: The Self-Report Habit Index (SRHI) will be used to assess habit formation. This index is a patient-reported outcome that examines habit strength. This self-report index comprises of 12 statements with constructs spanning behavior repetition, automaticity, and identity, with responses made on 11-point Likert scales (0 = strongly disagree; 10 = strongly agree). Higher scores indicate stronger habit formation (min = 0, max = 100).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percent (out of 100%)
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
percent (out of 100%) | 59.40 (26.57) | 44.08 (29.79)

13. Primary Outcome: Self-Report Habit Index (SRHI)
Description: as for outcome 12
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: percent (out of 100%)
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
percent (out of 100%) | 74.25 (20.72) | 57.85 (24.68)

14. Secondary Outcome: 10-Meter Walk Test (10MWT) - Comfortable Walking Speed
Description: This is a test of short-distance walking function. The participant will be asked to walk at comfortable walking speed (CWS) on a ten-meter straight walkway. Two trials will be administered, and the average of two trials will be reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 19
m/s | 1.16 (0.15) | 1.27 (0.16)

15. Secondary Outcome: 10-Meter Walk Test (10MWT) - Comfortable Walking Speed
Description: as for outcome 14
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 19
m/s | 1.18 (0.16) | 1.32 (0.15)

16. Secondary Outcome: 10-Meter Walk Test (10MWT) - Comfortable Walking Speed
Description: as for outcome 14
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 19
m/s | 1.18 (0.14) | 1.36 (0.16)

17. Secondary Outcome: 10-Meter Walk Test (10MWT) - Maximum Walking Speed
Description: This is a test of short-distance walking function. The participant will be asked to walk at maximum walking speed (MWS) on a ten-meter straight walkway. Two trials will be administered, and the average of two trials will be reported.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
m/s | 1.74 (0.36) | 1.82 (0.26)

18. Secondary Outcome: 10-Meter Walk Test (10MWT) - Maximum Walking Speed
Description: as for outcome 17
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
m/s | 1.77 (0.37) | 1.83 (0.32)

19. Secondary Outcome: 10-Meter Walk Test (10MWT) - Maximum Walking Speed
Description: as for outcome 17
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
m/s | 1.80 (0.36) | 1.80 (0.26)

20. Secondary Outcome: 6-Minute Walk Test (6MWT)
Description: This is test of long-distance walking function. The participant will be asked to "cover as much distance as they safely can" for 6 minutes, and total distance is the main metric from this test.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 19
m | 520.32 (86.99) | 548.56 (79.93)

21. Secondary Outcome: 6-Minute Walk Test (6MWT)
Description: as for outcome 20
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 19
m | 524.56 (83.56) | 562.31 (84.79)

22. Secondary Outcome: 6-Minute Walk Test (6MWT)
Description: as for outcome 20
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 20 | 19
m | 533.31 (92.65) | 570.98 (83.06)

23. Secondary Outcome: Gait Velocity During In-clinic Walking
Description: Quantified metrics of walking velocity (m/s) will be collected using wearable sensors.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 19 | 15
m/s | 1.50 (0.26) | 1.58 (0.22)

24. Secondary Outcome: Gait Velocity During In-clinic Walking
Description: Quantified metrics of walking velocity (m/s) will be collected using wearable sensors.
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 19 | 15
m/s | 1.53 (0.25) | 1.63 (0.25)

25. Secondary Outcome: Gait Velocity During In-clinic Walking
Description: Quantified metrics of walking velocity (m/s) will be collected using wearable sensors.
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 19 | 15
m/s | 1.55 (0.26) | 1.63 (0.25)

26. Secondary Outcome: Stride Length During In-clinic Walking
Description: Quantified metrics of stride length (m) will be collected using wearable sensors.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 19 | 15
m | 1.49 (0.18) | 1.54 (0.24)

27. Secondary Outcome: Stride Length During In-clinic Walking
Description: Quantified metrics of stride length (m) will be collected using wearable sensors.
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 19 | 15
m | 1.52 (0.20) | 1.56 (0.28)

28. Secondary Outcome: Stride Length During In-clinic Walking
Description: Quantified metrics of stride length (m) will be collected using wearable sensors.
Time Frame: Follow-up (up to 2 weeks post-intervention)
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 19 | 15
m | 1.53 (0.20) | 1.56 (0.25)

29. Secondary Outcome: Movement Disorder Society Unified Parkinson Disease Rating Scale Motor Subsection (MDS-UPDRS III)
Description: The MDS UPDRS is the most widely used clinical rating scale for Parkinson disease. Part III is a motor examination (33 scores summed from 18 questions) conducted by the rater. The total score is reported, which can range from 0 (no impairment) to 141 (maximum impairment).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 20.71 (7.68) | 22.75 (10.60)

30. Secondary Outcome: Movement Disorder Society Unified Parkinson Disease Rating Scale Motor Subsection (MDS-UPDRS III)
Description: as for outcome 29
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 23.48 (9.41) | 21.11 (18.74)

31. Secondary Outcome: Movement Disorder Society Unified Parkinson Disease Rating Scale Motor Subsection (MDS-UPDRS III)
Description: as for outcome 29
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 22.86 (10.15) | 18.74 (7.65)

32. Secondary Outcome: Self-Efficacy of Walking - Duration (SEW-D)
Description: The SEW-D is a 10-item self-report that will be administered to determine participants' beliefs of their physical capabilities to successfully complete incremental 5-minute intervals (5 to 40 minutes) of walking at a moderately fast pace, with responses made on 11-point Likert scale (0% = not at all confident; 100% = highly confident).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
percent | 73.76 (18.85) | 69.89 (18.83)

33. Secondary Outcome: Self-Efficacy of Walking - Duration (SEW-D)
Description: as for outcome 32
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
percent | 78.14 (19.49) | 76.95 (15.39)

34. Secondary Outcome: Self-Efficacy of Walking - Duration (SEW-D)
Description: as for outcome 32
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
percent | 78.57 (19.51) | 76.89 (19.48)

35. Secondary Outcome: Geriatric Depression Scale (GDS)
Description: The GDS is a brief, self-report involving yes/no questions instrument on psychological aspects and social consequences of depression in the elderly. The short form of GDS of 15-items will be used in this study. Higher scores indicate greater depression (min = 0, max = 15).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 2 (2.19) | 2.42 (2.34)

36. Secondary Outcome: Geriatric Depression Scale (GDS)
Description: as for outcome 35
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 2.24 (2.70) | 2.16 (2.09)

37. Secondary Outcome: Geriatric Depression Scale (GDS)
Description: as for outcome 35
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 2.76 (1.70) | 2.53 (1.54)

38. Secondary Outcome: Parkinson's Disease Questionnaire - 39 (PDQ-39)
Description: The PDQ- 39 is a self-report questionnaire that assesses quality of life over the past month across 8 different dimensions. Items are scored based on a 5-point ordinal system with lower scores reflecting better quality of life. Lower scores reflect better quality of life (min = 0, max = 100).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 11.95 (8.24) | 14.36 (8.46)

39. Secondary Outcome: Parkinson's Disease Questionnaire - 39 (PDQ-39)
Description: as for outcome 38
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 13.57 (8.92) | 15.44 (8.10)

40. Secondary Outcome: Parkinson's Disease Questionnaire - 39 (PDQ-39)
Description: as for outcome 38
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 12.34 (8.23) | 14.61 (9.23)

41. Secondary Outcome: Mini Balance Evaluation Systems Test (Mini BESTest)
Description: This test comprises of 14 items that span anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. Each item is scored from 0-2 (0 = lowest level of function, 2 = highest level of function). The total score is reported, calculated as the sum of all items, with possible scores of 0 (lowest level of balance function) and a maximum score of 28 (highest level of balance function).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 24.24 (2.43) | 24.89 (2.66)

42. Secondary Outcome: Mini Balance Evaluation Systems Test (Mini BESTest)
Description: as for outcome 41
Time Frame: Immediately after the intervention (up to 6 weeks)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 24.43 (2.09) | 25.84 (1.53)

43. Secondary Outcome: Mini Balance Evaluation Systems Test (Mini BESTest)
Description: as for outcome 41
Time Frame: Follow-up (up to 2 weeks post-intervention completion, and up to 8 weeks from baseline/start of intervention)
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Amped-PD | Active-Control
Number analyzed (Participants) | 21 | 19
points | 24.86 (2.03) | 26.00 (1.53)

ADVERSE EVENTS:
Time Frame: 8 weeks (includes 6-week intervention and 2-week follow-up)
Description: The 6-week walking program received by both intervention arms incurs negligible risk for all-cause mortality.
Arm/Group | Amped-PD | Active-Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 4/21 | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amped-PD (N=21) | Active-Control (N=20)
Fall (unrelated) (Nervous system disorders) | 2 (2) | 1 (1) — An unrelated fall is an unexpected, unplanned contact with a supporting surface that occurred outside of the walking program.
Fall (related) (General disorders) | 0 (0) | 2 (2) — A program-related fall is an unexpected and/ or unanticipated contact with the support surface while performing the walking program.
Toe pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Pain and soreness on toe, unrelated to the walking program.
Surgery (Hepatobiliary disorders) | 0 (0) | 1 (1) — Surgery involving gall bladder
Arm pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — General and non-specific report of pain on arm, unrelated to the walking program.
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) — Covid-19 infection with mild respiratory symptoms
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT05421624/Prot_004.pdf
  • Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT05421624/SAP_005.pdf
  • Informed Consent Form (2024-08-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT05421624/ICF_003.pdf